CLINICAL TRIAL: NCT06424314
Title: Changes in Respiratory Mechanics in Patients With Failed Ventilator Withdrawal
Brief Title: Exploration of Mechanisms for Weaning Failure
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Guan Lili, MD, The First Affiliated Hospital of Guangzhou Medical University
Other Study IDs: 202220252311
Record Dates: First submitted 2024-05-16; First posted 2024-05-22 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Weaning Failure; Central Respiratory Depression; Diaphragm Injury; Phrenic Nerve Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- weaning success: Patient passed SBT test with no need to receive invasive mechanical ventilation 48 hours after extubation
  Interventions: Diagnostic Test: Monitoring of respiratory mechanics parameters
- weaning failure: Patient failed SBT test or need to receive invasive mechanical ventilation 48 hours after extubation
  Interventions: Diagnostic Test: Monitoring of respiratory mechanics parameters

INTERVENTIONS:
Diagnostic Test: Monitoring of respiratory mechanics parameters — Physiologic recording instrumentation measure maximal transdiaphragmatic pressure，twitch diaphragmatic pressure and maximal diaphragmatic electromyography

SUMMARY:
This study is a prospective physiologic study. The primary study population will be adult invasive tracheal intubated patients with COPD, and investigators will collect relevant demographic data, vital signs, and baseline physiologic parameters of the patients prior to the spontaneous breathing test（SBT).

The participants will be divided into a successful withdrawal group and a failed withdrawal group according to the SBT outcome, and the changes in the above parameters during SBT will be compared between the two groups .

DETAILED DESCRIPTION:
This observational study mainly include participants who had invasive mechanical ventilation for ≥48 h and are assessed to be ready for the SBT trial.The SBT approach is based on the low-level pressure support mode.

Prior to the SBT trial, baseline demographic and physiologic data of the participants will be collected, and the participants will be divided into two groups based on the results of the SBT trial: successful and unsuccessful, and the physiologic changes during the SBT trial will be compared between the two groups, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Invasive mechanical ventilation for at least 48 hours

Exclusion Criteria:

* neuromuscular disease；Postoperative patients or patients with traumatic brain injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing weaning from mechanical ventilation；Hemodynamic stability
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
weaning success | Day 2
  passed SBT trial and weaning from mechanical ventilation success with no need of reintubation

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided